CLINICAL TRIAL: NCT05192083
Title: A Pilot Trial of a Smartphone-based Self-management Support Program for Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Pilot Trial of a Smartphone-based Self-management Support Program for COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW21-532-2
Record Dates: First submitted 2021-11-27; First posted 2022-01-14 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Self-management; Support; Smartphone-based
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Self-Management; Palliative Care

STUDY DESIGN:
Intervention Model Description: Self-management education and support
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The intervention group will receive a smartphone-based self-management support programme, including a 30-min face-to-face or online session at baseline, 3 phone calls (week 2, week 4 and week 6) and 2-month mobile messages in addition to usual care.
  Interventions: Behavioral: Self-management and Support

INTERVENTIONS:
Behavioral: Self-management and Support — A smartphone-based self-management support programme includes a 30-min face-to-face or online session at baseline, 3 phone calls and 2-month mobile messages

SUMMARY:
COPD patients often experience multiple symptoms (e.g. dyspnea, cough, and deteriorating quality of life) and have imposed a substantial economic and social burden on health care.

The current proposal is to evaluate the feasibility and acceptability of a pilot trial of a smartphone-based instant messaging self-management support program to improve the quality of life in patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the number 3 killer globally by 2020. COPD patients often experience multiple symptoms (e.g. dyspnea, cough, and deteriorating quality of life) and have imposed a substantial economic and social burden on health care.

Current policy for the prevention and management of long-term conditions focuses on efforts to prevent the onset or slow progression of disease early in the disease trajectory. This prevention paradigm has only recently been adopted for COPD. Systematic reviews have shown self-management support for patients with COPD is effective in improving health-related quality of life and in reducing hospital admissions, but the evidence comes largely from patients with moderate or severe disease and is predominantly recruited from secondary care. Simple and systematic strategies are needed to improve out-of-hospital support and management for people living with COPD.

An instant messaging smartphone app, which allows texts, audio, pictures and video messages to be shared in chat groups, is already available to and is the most popular in the Hong Kong general public. Mobile instant messaging can be conducted through a daily use device to increase access and efficacy, which has been suggested as a feasible approach to delivering an intervention with positive effects on health behaviours and outcomes. Text messaging via mobile phones has been shown to be effective in helping promote lifestyle change in diabetes self-management, weight loss, physical activity, smoking cessation and medication adherence with quantitative and qualitative evidence. However, the investigator has not found messaging intervention that was applied in people with COPD, except an ongoing study of using instant text message support for patients with chronic respiratory and cardiovascular diseases.

Hence, the current intervention program is to evaluate the feasibility and acceptability of a smartphone-based instant messaging self-management support program to improve the quality of life in patients with COPD.

ELIGIBILITY:
Inclusion criteria

* Aged 18 years and above
* Diagnosis with COPD
* General condition stable
* Able to speak and read Chinese
* Able to complete the self-administered questionnaire
* Able to use instant messages such as WhatsApp or WeChat
* Mental, cognitive and physically fit for joining the trial as determined by the clinician or responsible investigator
* Signed informed consent

Exclusion criteria

* Skeletal fragility
* Serious active infection
* Inability to walk
* Severe respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline COPD-related quality of life | Baseline, Week 8
  COPD symptoms and impacts and activity level were measured by an 8-item COPD Assessment Test. Total scores range from 0 to 40, with higher scores denoting a more severe impact of COPD on a patient's life.

SECONDARY OUTCOMES:
Change from baseline patient activation | Baseline, Week 8
  Knowledge, skills and confidence in self-management were measured by a 13-item Patient Activation Measure Scale. The total score ranges from 0 (no activation) to 100 (high activation), with higher scores denoting the better patient activation.
Change from baseline self-efficacy for self-management | Baseline, Week 8
  Confidence and perceived ability of self-care were measured by a 6-item Stanford self-efficacy scale. The score for each item ranges from 1 (not at all confident) to 10 (totally confident). The total score of the scale is the mean of the six items, with higher number indicates higher self-efficacy.
Change from baseline acceptance of illness | Baseline, Week 8
  Acceptance of illness measured by a 8-item acceptance of illness scale. Each item ranges from 1 to 5. The total score of the scale is between 8 and 40, with low score showing a lack of adjustment to the disease, no acceptance of the condition, and mental discomfort, while high score indicating good disease acceptance.
Change from baseline medication adherence | Baseline, Week 8
  Medication adherence measured by a 4-item Morisky Medication-Taking Adherence Scale. The scale consists of four items with a scoring scheme of "Yes" = 0 and "No" = 1. All items are summed to give a range of scores from 0 to 4, with higher score indicating a low level of medication adherence.
Change from baseline physical activity level | Baseline, Week 8
  Physical activity measured by a 7-item International Physical Activity Questionnaire-short form. Number of days and duration (in hours and minutes) engaging in vigorous activities, moderate activities, and walking in past 7 days will be collected. Duration (in hours and minutes) of sitting time on week days and weekends will be collected.
Change from dyspnea severity | Baseline, week 8
  Dyspnea severity measured by a 1-item MRC dyspnea scale. The scale consists of five statements about perceived breathlessness: grade 1, "I only get breathless with strenuous exercise"; grade 2, "I get short of breath when hurrying on the level or up a slight hill"; grade 3, "I walk slower than people of the same age on the level because of breathlessness or have to stop for breath when walking at my own pace on the level"; grade 4, "I stop for breath after walking 100 yards or after a few minutes on the level"; grade 5, " I am too breathless to leave the house". Patients selected the grade that applied to them.
Change from baseline Health status | Baseline, Week 8
  Health status measured by a 5-item EuroQol 5-Dimension questionnaire. The scale comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension was scored by five levels, with 1 representing no problem and 5 representing extreme problem.
Change from anxiety and depressive symptoms | Baseline, Week 8
  Anxiety and depressive symptoms measured by a 14-item Hospital Anxiety and Depression Scale. Each item ranges from 0-3. The total scores of both Anxiety and Depression subscales range from 0-21, with higher scores indicating higher level of anxiety and depression respectively.
Change in baseline social support | Baseline, Week 8
  Social support measured by a 6-item Multidimensional Scale of Perceived Social Support. Each item ranges from 1 (very strongly disagree) to 7 (very strongly agree). The total score is the sum across all items divided by 6, with higher score indicating more social support.
Change in from baseline sleep quality | Baseline, Week 8
  Sleep quality measured by a 7-item Insomnia Severity Index. The total score range from 0 (absence of insomnia) to 28 (severe insomnia).
Change in baseline grip strength | Baseline, Week 8
  Grip strength of both hands measured by dynamometer
Change in baseline balance | Baseline, Week 8
  Balance assessed by a single-leg stance test.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Need to obtain consent from patients before agreeing to share individual participants data.
Supporting Information: Study Protocol
Time Frame: When study finished
Access Criteria: The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Ms Asa Choi (email asachoi@hku.hk), (School of Nursing, The University of Hong Kong) for further information.

REFERENCES:
- [Background] Buttery SC, Zysman M, Vikjord SAA, Hopkinson NS, Jenkins C, Vanfleteren LEGW. Contemporary perspectives in COPD: Patient burden, the role of gender and trajectories of multimorbidity. Respirology. 2021 May;26(5):419-441. doi: 10.1111/resp.14032. Epub 2021 Mar 9. PMID 33751727
- [Background] Jolly K, Sidhu MS, Hewitt CA, Coventry PA, Daley A, Jordan R, Heneghan C, Singh S, Ives N, Adab P, Jowett S, Varghese J, Nunan D, Ahmed K, Dowson L, Fitzmaurice D. Self management of patients with mild COPD in primary care: randomised controlled trial. BMJ. 2018 Jun 13;361:k2241. doi: 10.1136/bmj.k2241. PMID 29899047
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- [Background] Redfern J, Hyun K, Singleton A, Hafiz N, Raeside R, Spencer L, Carr B, Caterson I, Cullen J, Ferry C, Santo K, Hayes A, Leung RWM, Raadsma S, Swinbourne J, Cho JG, King M, Roberts M, Kok C, Jenkins C, Chow C. ITM support for patients with chronic respiratory and cardiovascular diseases: a protocol for a randomised controlled trial. BMJ Open. 2019 Mar 1;9(3):e023863. doi: 10.1136/bmjopen-2018-023863. PMID 30826759
- See also: The top 10 causes of death — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death